CLINICAL TRIAL: NCT02121236
Title: Diagnostic Accuracy of Ultrasonography in Detecting Benign Radiolucent Lesions Compared to CBCT Imaging and Histological Examination
Brief Title: Diagnostic Accuracy of Ultrasonography in Detecting Benign Radiolucent Lesions
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-OraMed-02-2014
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Benign Radiolucent Lesions
Keywords: CBCT; Ultrasonic diagnosis; Benign radiolucent lesions; Histopathology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with benign radiolucent lesions

SUMMARY:
This is an in vivo study which aims to evaluate the diagnostic accuracy of ultrasonography in detecting benign radiolucent lesion in the both jaws. The ultrasonography-based diagnosis of contents will be compared to those findings obtained from the histological examination (i.e. the gold standard). The second part of this study will examine the measuring accuracy by comparing ultrasonography-based 3D measurements with those obtained from CBCT images of the lesion assuming that CBCT 3D measurements are the gold standard.

DETAILED DESCRIPTION:
Jaw is a common anatomical site for development of odontogenic and nonodontogenic lesions, and because of the wide variation of these lesions, the diagnosis is complex. Many techniques have been used to arrive at the final diagnosis such as conventional radiographs, computed tomography (CT), low dose cone beam CT, MRI.The use of ultrasonography has been shown to be important in evaluating the solid and cystic components of jaw lesions. Although ultrasound imaging technology is a safe and a minimally invasive procedure, and has been in use in medicine for many years, its use in dental medicine has been limited and mainly restricted to soft tissue applications. Studies evaluating the role of ultrasonography in the diagnosis of bone lesions of the jaw are limited.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a radiolucent or mixed-appearance intraosseous lesion in the upper or lower jaw requiring surgical removal
* no previous trauma to the maxillofacial region.
* no previous surgical intervention in the same area of the lesion.

Exclusion Criteria:

* the presence of a completely radiopaque lesion indicating solid content.
* patients with systemic conditions associated with bony pathology such as hyperparathyroidism, Paget disease, ﬁbrous dysplasia, multiple myeloma, etc...

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are primarily diagnosed as having a benign lesion in one of the two jaws are going to be included in the study. Patients are usually referred to the Oral and Maxillofacial Department at our University Dental School to confirm their primary diagnosis. A database of these referred patients will be created and a random sample from this database will be withdrawn.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Lesion Contents | One time assessment once sample recruitment has completed. Ultrasonographic images will be taken before the surgical intervention of the lesion, whereas the histological examination will be performed after the surgical removal
  Three possible categories for this variable: Solid, liquid, mixed.

SECONDARY OUTCOMES:
3D measurements of the lesion | One time assessment once sample recruitment has completed.

CONTACTS AND LOCATIONS:
Overall Officials: Obai Zainedeen, DDS MSc, Principal Investigator — PhD student, Department of Oral Medicine, University of Damascus Dental School, Damascus; Iyad Al-Haffar, DDS MSc Phd, Study Chair — Associate Professor of Oral Medicine, Department of Oral Medicine, University of Damascus Dental School, Damascus; Nabeel Kushaji, DDS MSc PhD, Study Director — Associate Professor of Oral Medicine, Department of Oral Medicine, University of Damascus Dental School
Locations (1):
- Department of Oral Medicine, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Lauria L, Curi MM, Chammas MC, Pinto DS, Torloni H. Ultrasonography evaluation of bone lesions of the jaw. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Sep;82(3):351-7. doi: 10.1016/s1079-2104(96)80365-9. PMID 8884838
- [Background] Abrahams JJ, Oliverio PJ. Odontogenic cysts: improved imaging with a dental CT software program. AJNR Am J Neuroradiol. 1993 Mar-Apr;14(2):367-74. PMID 8456714
- [Background] Mast HL, Haller JO, Solomon M. Benign lesions of the mandibular and maxillary region in children: characterization by CT and MRI. Comput Med Imaging Graph. 1992 Jan-Feb;16(1):1-9. doi: 10.1016/0895-6111(92)90193-d. PMID 1313327
- [Background] Tsiolis FI, Needleman IG, Griffiths GS. Periodontal ultrasonography. J Clin Periodontol. 2003 Oct;30(10):849-54. doi: 10.1034/j.1600-051x.2003.00380.x. PMID 14710764
- [Background] Imbeau J. Introduction to through-transmission alveolar ultrasonography (TAU) in dental medicine. Cranio. 2005 Apr;23(2):100-12. doi: 10.1179/crn.2005.015. PMID 15898566
- [Background] Gundappa M, Ng SY, Whaites EJ. Comparison of ultrasound, digital and conventional radiography in differentiating periapical lesions. Dentomaxillofac Radiol. 2006 Sep;35(5):326-33. doi: 10.1259/dmfr/60326577. PMID 16940480